CLINICAL TRIAL: NCT04506580
Title: Comparison of Postoperative Wound Between Dermabond PRINEO™(2-octyl Cyanoacrylate Adhesive and Polyester Mesh) and Subcuticular Suture in Simultaneous Total Knee Arthroplasty
Brief Title: Comparison of Postoperative Wound Between Dermabond Prineo(2-octyl Cyanoacrylate Adhesive and Polyester Mesh) and Subcuticular Suture in Simultaneous Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Head of Orthopaedic Surgery, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dermabond vs. Subcuticular
Record Dates: First submitted 2020-02-01; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Knee Cutaneous Suture, Dermabond, Subcuticular Suture
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermabond group (Experimental): close capsule using 1-0 vicryl suture material close subq layer using 1-0 and 2-0 bicryl suture material and close skin layer using DERMABOND™ PRINEO™
  Interventions: Procedure: DERMABOND™ PRINEO™(2-octyl Cyanoacrylate Adhesive and Polyester Mesh) vs subcuticular nylon suture
- Subcuticular group (No Intervention): close capsule using 1-0 vicryl suture material close subq layer using 1-0 and 2-0 bicryl suture material and close skin layer using 3-0 Dermalon with subcuticular suture method

INTERVENTIONS:
Procedure: DERMABOND™ PRINEO™(2-octyl Cyanoacrylate Adhesive and Polyester Mesh) vs subcuticular nylon suture — DERMABOND™ PRINEO™(2-octyl Cyanoacrylate Adhesive and Polyester Mesh) and subcuticular nylon suture are applied for each knee
  Arms: Dermabond group

SUMMARY:
This study aims to compare the clinical results of postoperative wound between Dermabond PRINEO™(2-octyl Cyanoacrylate adhesive and polyester mesh) and subcuticular suture in simultaneous total knee arthroplasty

There is previous studies over whether or not to use skin adhesive material is superior or inferior to subcuticular suture This study prospectively randomized patients receiving bilateral total knee arthroplasty(TKA). Patients preference and clinical results was investigated in both knee of same patients who received skin adhesive or subcuticular suture in each knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty
* having medicare insurance

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Allergy or intolerance to study material
* Patients with an American Society of Anesthesiologists(ASA) score of IV (angina, congestive heart failure, dementia, cerebrovascular accident)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
wound Hypertrophy scale at postoperative 6 month | at postoperative 6 months
  Vancouver scar scale, patient and observer report scar assessment scale

SECONDARY OUTCOMES:
Skin closure time | operation day
  Skin closure time for each group
wound complication | postoperative 2 weeks
wound complication | postoperative 6 weeks
wound complication | postoperative 3 month
wound complication | postoperative 6 month
Stitch out time | postoperative 2 weeks
Stitch out visual visual analogue scale(VAS) | postoperative 2 weeks
  VAS range from 1 to 10 ( 1means minimal pain 10 means maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Study Chair — the Catholic Univerisity of Korea Seoul St Mary's hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No